CLINICAL TRIAL: NCT04880785
Title: Virologic Outcomes of Lamivudine/Dolutegravir in Virologically Suppressed Subjects With Expected or Confirmed Resistance to Lamivudine.
Brief Title: Lamivudine/Dolutegravir in Virologically Suppressed Subjects With Expected or Confirmed Resistance to Lamivudine
Acronym: VOLVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA11820
Record Dates: First submitted 2021-04-29; First posted 2021-05-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Lamivudine; Tablets

STUDY DESIGN:
Intervention Model Description: Phase IIa, open-label, single arm, multicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dovato (Dolutegravir+lamivudine) (Experimental): Treatment: Dolutegravir 50 mg/Lamivudine 300 mg, one film coated-tablet once daily during 96 weeks
  Interventions: Drug: Dolutegravir 50 MG / Lamivudine 300 MG Oral Tablet [Dovato]

INTERVENTIONS:
Drug: Dolutegravir 50 MG / Lamivudine 300 MG Oral Tablet [Dovato] — change of current antiretroviral treatment to DTG 50 mg/3TC 300 mg QD

SUMMARY:
Dolutegravir (DTG) plus lamivudine (3TC) is a dual regimen combination recommended for both naïve and suppressed persons with HIV-1 infection1. However, data regarding the efficacy of this regimen in suppressed persons with history of past resistance or virologic failures is currently insufficient. This is a phase IIa, open-label, single arm, multicentric study.

The hypothesis is that therapy with DTG/3TC would be able to maintain viral control in HIV infected participants with prior history of 3TC resistance but without evidence of M184V/I resistance mutation in proviral DNA population sequencing at baseline. The investigators also hypothesize that archived minority 3TC resistance associated mutations detected by next-generation (NGS) sequencing prior to the switch would not have a significant impact on the efficacy of DTG/3TC.

DETAILED DESCRIPTION:
This is a multicentre study, and it will be conducted at different healthcare centres in Spain. 117 participants will be recruited. A minimum of 30%-50% of the study population would be required to have historical RNA population genotype with confirmed M184V/I mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>=18 years old) with HIV-1 infection able to understand and give informed written consent.
2. Stable ART in the 12 weeks prior to screening visit.

   - Only switch for tolerability/convenience/access reasons to generic drugs or switch from ritonavir to cobicistat or TDF to TAF would be allowed in the 12-week window and as long as the components of the regimen are unchanged.
3. Viral load <50 copies/mL at screening and in the year prior to study entry.

   - A blip (50-500 copies/ml) would be allowed within 48 weeks prior to inclusion in the study, if preceded and followed by an undetectable VL determination.
4. CD4 count > 200 cel/μL at screening.
5. History of 3TC resistance: either confirmed historical 3TC resistance (historical RNA Sanger or RNA NGS>20% threshold genotype with M184V/I mutation) OR suspected historical 3TC resistance.

   * Suspicion of past 3TC resistance is defined as any of the following:

i. Previous treatment with only 2 NRTIs (1 of them being emtricitabine or 3TC [XTC]).

ii. Two consecutive VL > 200 cp/mL while on treatment including XTC. iii. One VL > 200 cp/mL while on treatment including XTC PLUS change of ART as consequence of that elevated VL.

Exclusion Criteria:

1. Participants with M184V/I or K65R in screening visit proviral DNA Sanger genotype.
2. Prior virologic failure (VF) under integrase inhibitor (INSTI)- based regimen. defined as two consecutive VL > 200 copies/mL while receiving INSTI regardless of genotypic test results
3. INSTI resistance mutations in historical RNA genotype.
4. Positive Surface Hepatitis B Ag (HBAgS) OR negative HBAgS and negative hepatitis B surface antibody (anti-HBs) with positive anti-core antibody (anti-HBc) and positive HBV DNA.
5. Pregnant, breastfeeding women, women with a positive pregnancy test at the time of screening, sexually active fertile women wishing to conceive or unwilling to commit to contraceptive methods (see Appendix 1 for the accepted list of the highly effective methods for avoiding pregnancy), for the duration of the study and until 4 weeks after the last dose of study medication. All women are considered fertile unless they have undergone a sterilizing surgery or are over the age of 50 with spontaneous amenorrhea for over 12 months prior to study entry.
6. Patients with active opportunistic infections or cancer requiring intravenous treatment and/or chemotherapy at screening.
7. Any comorbidities or treatment with experimental drugs that according to the investigator could bias study results or entail additional risks for the participant.
8. Participants receiving other medications that according to study drug label are contraindicated.
9. Severe hepatic impairment (Class C) as determined by Child-Pugh classification.
10. Alanine aminotransferase (ALT) over 5 times the upper limit of normal (ULN) or ALT over 3xULN and bilirubin over 1.5xULN.
11. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (apart from hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones);
12. Creatinine clearance of <30 mL/min/1.73m2 via CKD-EPI method.
13. Any verified Grade 4 laboratory abnormality that to the investigators criteria would affect the safety of the participant if included in the study.
14. History or presence of allergy to dolutegravir or lamivudine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
The efficacy of a switch to DTG/3TC for maintenance of virologic suppression, in persons with past confirmed or suspected 3TC resistance, when proviral DNA population sequencing does not detect 3TC resistance-associated mutations at baseline. | Week 48
  Proportion of virologic failure (VF) defined as HIV-1 RNA viral load (VL) ≥ 50 copies per mL (in the intention-to-treatexposed population (ITT-e) using the US Food and Drug Administration (FDA) snapshot algorithm).

SECONDARY OUTCOMES:
Estimations of virological control | Week 48 and week 96
  Proportion of VF (≥50 copies/mL) ITT-e, per protocol population (PP), Proportion of VF (≥200 copies/mL), ITT-e and PP population, FDA snapshot. Proportion of Confirmed Virologic Withdrawal ([CVW]: A VL≥ 50 copies/mL followed by a VL≥ 200 copies/mL in retest), ITT-e and PP population, FDA snapshot. Proportion of Precautionary Virologic Withdrawal ([PVW]: three consecutive VL between 50- 200 copies/mL), ITT-e and PP population, FDA snapshot. Proportion of participants with VL<50 copies/mL, ITT-e and per protocol population, FDA snapshot.
Viral resistance in persons experiencing VF. | Throughout all the study, an average of 96 weeks
  Incidence of VF with drug resistance associated mutations.
  - Describe number and type of resistanceassociated mutations in VF
Time to VF | Throughout all the study, an average of 96 weeks
Proportion of VF in subgroups: Confirmed historical M184V/I vs No resistance mutations | Throughout all the study, an average of 96 weeks
Proportion of VF in subgroups: INSTI exposure vs No prior INSTI exposure | Throughout all the study, an average of 96 weeks
Time virologically suppressed | Throughout all the study, an average of 96 weeks
Proportion of VF in subgroup: Time on 3TC/FTC | Throughout all the study, an average of 96 weeks
Proportion of participants with VF with baseline 3TC or INSTI resistanceassociated mutations detected at baseline by NGS with 1, 5, and 20% threshold. | Throughout all the study, an average of 96 weeks
  Proportion of participants with transient viral rebounds with baseline 3TC or INSTI resistance- associated mutations detected at baseline by NGS with 1, 5, and 20% threshold.
Proportion of participants with transient viral rebounds with baseline 3TC or INSTI resistance- associated mutations detected at baseline by NGS with 1, 5, and 20% threshold. | Throughout all the study, an average of 96 weeks
Type of resistance mutations (RT and integrase) in proviral DNA measured by NGS. | Throughout all the study, an average of 96 weeks
Frequency of resistance mutations (RT and integrase) in proviral DNA measured by NGS. | Throughout all the study, an average of 96 weeks
Change in CD4+ cell count | Basal, Week 48 and week 96
Change in CD4+/CD8+ cell counts ratio | Basal, Week 48 and week 96
Incidence and severity of AEs and laboratory abnormalities. | Basal, Week 48 and week 96
Proportion of subjects who discontinue treatment due to AEs | Basal, week 48 and week 96

CONTACTS AND LOCATIONS:
Locations (17):
- Spain (17):
  - H. Álvaro Cunqueiro, Vigo, Pontevedra
  - CHUAC, A Coruña
  - H. de Elche, Alicante
  - H. General de Alicante, Alicante
  - H. Bellvitge, Barcelona
  - H. Clinic, Barcelona
  - H. del Mar, Barcelona
  - H. de Donosti, Donostia / San Sebastian
  - H. Fundación Jimenez Díaz, Madrid
  - H. Infanta Leonor, Madrid
  - H. La Princesa, Madrid
  - H. Príncipe de Asturias, Madrid
  - H. Severo Ochoa, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital General Univ. Gregorio Marañón, Madrid
  - Hospital Univ. La Paz, Madrid
  - H. Virgen de la Victoria, Málaga

DOCUMENTS (1):
  • Study Protocol (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT04880785/Prot_000.pdf